CLINICAL TRIAL: NCT06515184
Title: Coenzyme Q10 for Gulf War Illness: A Replication Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Beatrice Golomb, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GW190064
Record Dates: First submitted 2024-06-10; First posted 2024-07-23 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Gulf War Syndrome; Persian Gulf Syndrome; Mitochondrial Disorder, Respiratory Chain
MeSH Terms: conditions — Persian Gulf Syndrome; Mitochondrial Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Design (primary) is followed by active treatment phase (still blind to dose).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CoQ10 Arm 1 (Active Comparator): PharmaNord Ubiquinone 100mg/1x day
  Interventions: Drug: PharmaNord Bio-Quinone Active CoQ10 Gold 100mg
- CoQ10 Arm 2 (Active Comparator): PharmaNord Ubiquinone 100mg/3x day
  Interventions: Drug: PharmaNord Bio-Quinone Active CoQ10 Gold 100mg
- Placebo Arm (Placebo Comparator): Placebo (made by PharmaNord, matches active treatment)
  Interventions: Drug: PharmaNord Placebo

INTERVENTIONS:
Drug: PharmaNord Bio-Quinone Active CoQ10 Gold 100mg — Each participant receives one softgel three times a day. Arm 1 receives one 100mg softgel and two placebo softgels per day.
  Because of the presence of the IND, the dropdown menu does not allow us to choose dietary supplement. The option "drug" was chosen as the closest permissible option.
  Arms: CoQ10 Arm 1
Drug: PharmaNord Placebo — Each participant receives one softgel three times a day. Arm 3 receives three placebo softgels per day. Supplement is taken orally in divided doses, with the last softgel not close to bedtime.
  Because of the presence of the IND, the dropdown menu does not allow us to choose dietary supplement. The option "drug" was chosen as the closest permissible option.
  Arms: Placebo Arm
Drug: PharmaNord Bio-Quinone Active CoQ10 Gold 100mg — Each participant receives one softgel three times a day. Arm 2 receives three 100mg softgels per day. Supplement is taken orally in divided doses, with the last softgel not close to bedtime.
  Because of the presence of the IND, the dropdown menu does not allow us to choose dietary supplement. The option "drug" was chosen as the closest permissible option.
  Arms: CoQ10 Arm 2

SUMMARY:
The purpose of this study is to assess whether a high quality preparation of ubiquinone (coenzyme Q10) benefits symptoms, function, and quality of life in veterans with Gulf War illness.

ELIGIBILITY:
Inclusion Criteria:

* Meets both CDC and Kansas deployment and symptom inclusion criteria.
* Does not have a disqualifying condition.
* Able to travel to a local Quest facility for study blood draws.
* Adequate internet access to allow ZoomPro visit participation and remote survey completion.
* Health prior to the Gulf War rated as "very good" or "excellent" (to exclude persons who may have had other health conditions with different mechanisms as the cause of their symptoms).
* Willing to defer initiation of discretionary treatments or supplements during the expected course of study participation.

Exclusion Criteria:

* Participating in another clinical trial.
* Still-evolving adverse effects following another medication or health condition, such as covid or fluoroquinolone use.
* On Coumadin/ warfarin.
* Unable to participate for the required duration of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of symptoms (out of 20 on the UCSD Symptom Score Survey) showing more favorable change (trend or effect) on active treatment vs. on placebo. | 3.5 months
  All outcomes are assessed as change from baseline.

SECONDARY OUTCOMES:
Percent improved on timed chair rises from Gulf War Illness Modified Lower Extremity Summary Performance Score. | 3.5 months
  All outcomes are assessed as change from baseline.
Mean change in single-item General Self-Rated Health (GSRH). | 3.5 months
  All outcomes are assessed as change from baseline. 5 point scale, higher is good.
Individual GWI Symptoms | 3.5, 7 months
  7 validated single-item symptom self-ratings: headache; energy; fatigue with exertion, muscle pain; irritability; impatience; trouble recalling words/names. Each benefited with coQ10, p<0.05 (two-sided), in the prior coQ10 trial.
Relation of change in time to do five chair rises to change in blood level of coenzyme Q10 | 3.5, 7 months
  Benefit to timed chair rises will relate to blood coQ10 change. This outcome assesses the relation between change in time to complete five chair rises (in seconds) to change in blood level of CoQ10 (in ug/mL). The prediction of change in time to perform five chair rises by change in coQ10 blood level (regression with robust standard errors).
Effect of CoQ10 in the majority male subset on symptoms. | 3.5, 7 months
  Change in symptoms on coQ10 versus placebo will be assessed in men (male subset of sample).
Effect of CoQ10 in the majority male subset on timed chair rises. | 3.5, 7 months
  Change in timed chair rises on coQ10 versus placebo will be assessed in men (male subset of sample).
Effect of CoQ10 in the majority male subset on GSRH. | 3.5, 7 months
  Change in GSRH on coQ10 versus placebo will be assessed in men (male subset of sample).

OTHER OUTCOMES:
The investigator will assess whether there is a difference in change effect for the 100mg/day vs 300mg/day arm on symptoms. | 3.5, 7 months
  Compare the effect of coQ10 300mg/day to placebo, and to coQ10 100mg/d on symptoms.
The investigator will assess whether there is a difference in change effect for the 100mg/day vs 300mg/day arm on timed chair rises. | 3.5, 7 months
  Compare the effect of coQ10 300mg/day to placebo, and to coQ10 100mg/d on timed chair rises.
The investigator will assess whether there is a difference in change effect for the 100mg/day vs 300mg/day arm on GSRH. | 3.5, 7 months
  Compare the effect of coQ10 300mg/day to placebo, and to coQ10 100mg/d on GSRH.
Duration Effect on symptoms. Compare effects of 7 months vs 3.5 months of treatment, assessed at the same time point after baseline (7 months) on symptoms. | 7 months
  Following seven months of study participation, participants will have been on coQ10 for either 3.5 months or 7 months. These two groups will be compared to assess the impact of longer vs. shorter duration treatment (those initially randomized to placebo will crossover to active coQ10 for the final 3.5 months, while those originally randomized to coQ10 will have been on coQ10 for 7 months).
Duration Effect on timed chair rises. Compare effects of 7 months vs 3.5 months of treatment, assessed at the same time point after baseline (7 months) on timed chair rises. | 7 months
  Following seven months of study participation, participants will have been on coQ10 for either 3.5 months or 7 months. These two groups will be compared to assess the impact of longer vs. shorter duration treatment (those initially randomized to placebo will crossover to active coQ10 for the final 3.5 months, while those originally randomized to coQ10 will have been on coQ10 for 7 months).
Duration Effect on GSRH. Compare effects of 7 months vs 3.5 months of treatment, assessed at the same time point after baseline (7 months) on GSRH. | 7 months
  Following seven months of study participation, participants will have been on coQ10 for either 3.5 months or 7 months. These two groups will be compared to assess the impact of longer vs. shorter duration treatment (those initially randomized to placebo will crossover to active coQ10 for the final 3.5 months, while those originally randomized to coQ10 will have been on coQ10 for 7 months).
Blood Pressure | 3.5, 7 months
  Specifically, change in blood pressure on coq10 versus placebo will be assessed considering those with low blood pressure at baseline separately from those with borderline or high blood pressure at baseline.
Mitochondrial Function from blood spot card. Maximal respiration will be assessed by the "adopted transfer" technique. | 3.5, 7 months
Mitochondrial Function from blood spot card. Spare capacity will be assessed by the "adopted transfer" technique. | 3.5, 7 months
Inflammation (hsCRP) will be assessed as change from baseline and compared on active treatment vs. placebo. | 3.5, 7 months
Oxidative Stress | 3.5, 7 months
Liver Function. Alanine aminotransferase and aspartate aminotransferase will be assessed as change from baseline and compared on active treatment vs. placebo. | 3.5, 7 months
Dropouts for Cause. The investigator will report participants who drop out for a reason. | 3.5, 7 months
  For instance, participants who transition from coQ10 to placebo might drop because of lost of needed benefits of coQ10 -- because the participant felt worse. Alternatively, participants who transition from placebo run-in to coQ10 might drop out due to problems like activation insomnia on active treatment. The number of dropouts will be compared on active treatment vs placebo, and the causes of dropout will be compared also. (Participants who drop because their physicians ask them to do so for some unrelated reason, not because the patient has had a problem or perceive a problem, will count as dropouts, but not as dropouts for "cause" -- cause here refers to a symptom change and/or medical event.) In addition to overall assessment, assessment of dropouts for cause will be evaluated stratified by whether the participant is transitioning from coQ10.
Relation of change in symptoms to change in blood level of coenzyme Q10 | 3.5 +/- 0.5 months (priority), and ~7 months
  This outcome assesses the relation between change in symptoms to change in blood level of CoQ10 (in ug/mL).
Relation of change in single-item General Self-Rated Health (GSRH) to change in blood level of coenzyme Q10 | 3.5, 7 months
  This outcome assesses the relation between change in single-item General Self-Rated Health (GSRH) to change in blood level of CoQ10 (in ug/mL). The GSRH is a 5 point scale, higher is good.
Subset effects in those citing prior coQ10 use, stratified by whether benefit had been perceived. | 3.5, 7 months
Analysis stratified by presence of symptoms compatible with sleep apnea | 3.5, 7 months
  For inclusion in sleep apnea stratum during analysis, the following will be qualifying: Diagnosed sleep apnea, nocturia, awaking from sleep gasping or choking (or observed by others gasping or choking during sleep), daytime hypersomnolence, night sweats, or awaking with headache or anxiety. This is exploratory, but each outcome will be stratified by sleep apnea-compatible problems.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice A Golomb, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-09-12): https://cdn.clinicaltrials.gov/large-docs/84/NCT06515184/ICF_001.pdf